CLINICAL TRIAL: NCT01868607
Title: Comparison of the Reliability of Different Devices to Measure Lung Function With the Forced Oscillation Technique
Brief Title: Reliability of Different FOT Devices to Measure the Human Respiratory Impedance
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Ellie Oostveen, Professor Ellie Oostveen, University Hospital, Antwerp
Other Study IDs: FOT_UZA_2013
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Pulmonary Disease; Healthy
Keywords: Respiratory resistance; Respiratory reactance; Adult lung function; Forced oscillation technique; subjects
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult lung function

SUMMARY:
The objective of the study is to evaluate the reliability of the impedance data in adult subjects measured with five different FOT devices.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the reliability of the respiratory impedance measured with different FOT (=Forced Oscillation Technique) devices. To this end, the respiratory impedance of fifty adult subjects will be measured in random order with five different forced oscillation devices. As there is no "gold standard" FOT-device, each setup will be compared to all other setups.

Secondary study questions are: 1) is there a specific comfort (or discomfort) associated with the different measuring devices 2) Guidelines state that full chin and cheek support should be applied when measuring the human respiratory impedance. What is the influence of a partial cheek support?

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects
* Adult patients with obstructive lung disease

Exclusion Criteria:

* Inability to perform lung function tests
* Patients with respiratory failure
* Patients on BIPAP-therapy
* Patients on supplemental oxygen.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult subjects and patients with obstructibve lung disease
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the respiratory impedance measured with two different FOT devices | 1 day
  Bland-Altman plot of Zrs measured with two devices

SECONDARY OUTCOMES:
Subjective evaluation of the Zrs-measurement with a specific FOT device by the investigated subject. | 1 day
  Rating of the subjective experience of the Zrs-measurement with a specific FOT device

OTHER OUTCOMES:
Effect of the mode of cheek support on the Zrs-measurement | 1 day
  The effect of two modes of cheek support on the Zrs-estimate will be assessed in each investigated subject with one (randomly chosen) FOT-device.

CONTACTS AND LOCATIONS:
Overall Officials: Ellie Oostveen, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Dept. of Pulmonary Medicine, Antwerp University Hospital, Edegem-Antwerp, Belgium

REFERENCES:
- [Background] Oostveen E, MacLeod D, Lorino H, Farre R, Hantos Z, Desager K, Marchal F; ERS Task Force on Respiratory Impedance Measurements. The forced oscillation technique in clinical practice: methodology, recommendations and future developments. Eur Respir J. 2003 Dec;22(6):1026-41. doi: 10.1183/09031936.03.00089403. PMID 14680096
- [Background] Oostveen E, Boda K, van der Grinten CP, James AL, Young S, Nieland H, Hantos Z. Respiratory impedance in healthy subjects: baseline values and bronchodilator response. Eur Respir J. 2013 Dec;42(6):1513-23. doi: 10.1183/09031936.00126212. Epub 2013 Apr 18. PMID 23598954
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172